CLINICAL TRIAL: NCT01894438
Title: Effect of a Mediterranean Lifestyle Intervention on Biochemical and Clinical Characteristics of Patients With Non-alcoholic Fatty Liver Disease.
Brief Title: Mediterranean Lifestyle Intervention in Patients With Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Collaborators: University of Athens (Other)
Responsible Party: Principal Investigator, Meropi Kontogianni, Lecturer of Clinical Nutrition, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LD-0098
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD); Non-alcoholic Steatohepatitis (NASH)
Keywords: NAFLD; NASH; Mediterranean diet; Mediterranean lifestyle
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Diet, Mediterranean

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Group (No Intervention): This arm will receive written general advice for a healthy lifestyle.
- Mediterranean Diet Group (Experimental): Mediterranean Diet Group participants will attend a comprehensive program,focusing on Mediterranean diet, comprising of seven 60-min group counseling sessions, conducted every two weeks for the first 2 months and every month for the following 4 months, until the 6-month evaluation.
  Interventions: Behavioral: Mediterranean Diet
- Mediterranean Lifestyle Group (Experimental): Mediterranean Lifestyle Group participants will attend a comprehensive program,focusing on Mediterranean lifestyle, comprising of seven 60-min group counseling sessions, conducted every two weeks for the first 2 months and every month for the following 4 months, until the 6-month evaluation.
  Interventions: Behavioral: Mediterranean lifestyle

INTERVENTIONS:
Behavioral: Mediterranean lifestyle — Counseling will be based on the goal setting theory. Motivational and behavioral strategies will be also used. In the Mediterranean lifestyle group culinary practices, seasonality, and locality of food products, socialization during meals, rest during the day, as well as the adoption of an active living will be additionally addressed.
  Arms: Mediterranean Lifestyle Group
Behavioral: Mediterranean Diet — Counseling will be based on the goal setting theory. Motivational and behavioral strategies will be also used. In the Mediterranean diet group, all food groups of the Mediterranean diet will be targeted.
  Arms: Mediterranean Diet Group

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is considered as the hepatic manifestation of the metabolic syndrome. NAFLD is a pathologic condition which involves both hepatic steatosis and non alcoholic steatohepatitis (NASH), as the result of fat accumulation in the liver (liver fat >5-10% of liver weight), not due to excess alcohol consumption or other causes of steatosis.

At present, no medication or surgical procedure has been approved for treating NAFLD and lifestyle modifications remain the cornerstone therapy targeting both at weight reduction for overweight subjects and at prevention of overweight for the normal weight individuals. Given that a Mediterranean dietary pattern has a beneficial effect both on the prevention and the resolution of the metabolic syndrome, the main aim of the present study is to implement and evaluate the potential benefits of an intervention based on the Mediterranean lifestyle in a sample of patients with NAFLD.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is a pathologic condition which involves both hepatic steatosis and non alcoholic steatohepatitis (NASH), as the result of fat accumulation in the liver (liver fat >5-10% of liver weight), not due to excess alcohol consumption or other causes of steatosis. Its prevalence ranges in the general population from 10-35%, while in obese individuals can reach the 75% and is particularly worrying because these people appear to have a higher mortality from both liver and non-liver-related disease, such as cardiovascular disease, and therefore a greater economic burden of health costs.

At present, no medication or surgical procedure has been approved for treating NAFLD and lifestyle modifications remain the cornerstone therapy targeting both at weight reduction for overweight subjects and at prevention of overweight for the normal weight individuals. Given that a Mediterranean dietary pattern has a beneficial effect both on the prevention and the resolution of the metabolic syndrome, the main aim of the present study is to implement and evaluate the potential benefits of an intervention based on the Mediterranean lifestyle in a sample of patients with NAFLD. A secondary aim will be to produce material, for both health professionals (namely dietitians and doctors) and patients to help them implementing such an intervention based on the Mediterranean lifestyle.

This study will be a prospective, randomized, blinded and controlled study. Participants with NAFLD and BMI>25Kg/m2 (range 25-40 Kg/m2) will be included. NAFLD's diagnosis will be based on increased serum levels of alanine aminotransferase (ALT), with or without increased gamma-glutamyl transpeptidase (GGT) serum levels, the presence of hepatic steatosis and absence of other causes of hepatic steatosis and hepatic failure.

At baseline, patients will be informed about the study and will give their written consent. Then subjects will be randomly assigned to one of 3 groups: (a) Control group, receiving written general advice for a healthy lifestyle; (b) Mediterranean diet Group or (c) Mediterranean lifestyle group. Participants in (b) and (c) groups will attend a more comprehensive program, comprising seven 60-min group counseling sessions, conducted every two weeks for the first 2 months and every month for the following 4 months, until the 6-month evaluation. Participants will be also assessed 12 months after their entry in the study.

The dietary intervention and the monitoring will be carried out in the laboratory of Clinical Nutrition & Dietetics at Harokopio University, where experienced clinical dietitians will conduct all consultations. Counseling will be based on the goal setting theory. Motivational and behavioral strategies will be also used. In the Mediterranean diet group, all food groups of the Mediterranean diet will be targeted, whereas in the Mediterranean lifestyle group culinary practices, seasonality, and locality of food products, socialization during meals, rest during the day, as well as the adoption of an active living will be additionally addressed. Intervention will also aim at achieving a 5-10% weight loss within the first 6 months.

Patients will be evaluated at baseline, at the end of the 6-mo intervention and 1 year after the study entry. At baseline, all patients will undergo a brief medical history assessment, complete physical examination and routine laboratory testing. History of alcohol consumption will be obtained from both patients and friends/relatives where possible. Evaluation of anthropometric measurements, dietary intake, physical activity and lifestyle habits, will be continuously assessed throughout the study. Dietary intake will be assessed through two 24-hour recalls and a food frequency questionnaire (FFQ). Data from recalls will be analyzed in terms of energy, macro- and micronutrient intake (using the Nutritionist Pro, version 2.2 software), as well as of food group intake and meal patterns. Conditions around eating will be also recorded and analyzed. Furthermore, a semi-quantitative FFQ, including the main food groups of the Mediterranean diet will be used for the overall assessment of eating habits. Physical activity will be assessed using the Harokopio Physical Activity Questionnaire (HPAQ). Sleep duration and quality will be evaluated through the Athens Insomnia Scale, consisting of items related to sleep induction, awakenings during the night, final awakening, total sleep duration, and sleep quality, well-being, functioning capacity, and sleepiness during the day. Current and past smoking habits will be also recorded.

At baseline and at 6 and 12 months, blood samples will be collected after an overnight food deprivation for the assessment of biochemical markers, and stored at -80oC. Lipid profile, markers of glucose metabolism and liver function, and adipokines, inflammatory markers and markers of oxidative stress will be determined using automated analyzers and/or commercial ELISA kits.

All patients will pass through liver stiffness measurements with liver elastography at baseline, as well as at the end of the intervention and after one year of the study entry. Patients without a recent liver biopsy (within the previous 12 months) will also undergo liver biopsy at baseline. Liver biopsies will be repeated one year after and will be evaluated by the same hepato-pathologist, who will have access to patient's clinical data.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria will be:

* Participants aged 18-65 years old,
* Participants with non-alcoholic fatty liver disease (NAFLD). NAFLD's diagnosis will be based on increased serum levels of alanine aminotransferase (ALT) above 1.5 times, with or without increased gamma-glutamyl transpeptidase (GGT) serum levels,
* BMI >25 Kg/m2 (range 25-40 Kg/m2),
* The presence of hepatic steatosis and absence of other causes of hepatic steatosis and hepatic failure.

Exclusion Criteria:

The exclusion criteria will be:

* Detection of hepatitis B surface antigen (HBsAg) or antibodies against hepatitis C(anti-HCV) or antibodies against HIV,
* Alcohol intake >210 or >140 gr per week for men or women, respectively,
* Reception of potentially hepatotoxic drugs,
* Presence of systemic disease with potential liver involvement,
* Diabetes mellitus.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-04; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Serum levels of alanine aminotransferase (ALT) | Within 6 months
  Clinically useful reduction in ALT, defined as the restoration of ALT within normal limits or reduction of ALT in >50% of its initial value.

SECONDARY OUTCOMES:
Gamma-glutamyl transpeptidase (GGT) | Within 6 months
  Restore of GGT levels within normal limits (i.e. GGT<30 IU/L).
Liver stiffness | Within 6 months
  Improved liver stiffness as estimated with elastography.
Inflammatory and oxidative stress markers | Within 6 months
  Improved inflammatory markers (TNF-a, IL-6, IL-8, adiponectin) and oxidative stress markers (ex vivo serum resistance to oxidation, measurement of the compounds that react with thiobarbituric acid-TBARS, activity of glutathione peroxidase) as well as lipid/glucose metabolism improvement (triglycerides, HDL, LDL, total cholesterol, insulin resistance index).

CONTACTS AND LOCATIONS:
Overall Officials: Meropi D. Kontogianni, PhD, Study Director — Harokopio University
Locations (1):
- Harokopio University, Kallithea, Attica, Greece

IPD SHARING:
Plan to Share IPD: No
Data will be available upon demand.